CLINICAL TRIAL: NCT03298568
Title: Pilotstudie Zur Untersuchung Der Wirkung Einer Oralen Supplementation Von Diaminooxidase (DAOsin®) Bei Histamin-Intoleranz in Bezug Auf Die Steigerung Der Erniedrigten Endogenen Diaminooxidase-Aktivität
Brief Title: Study to Investigate the Effect of an Oral Diamine Oxidase Substitution (DAOsin) in Histamine Intolerant Patients on the Low Endogenous Diamine Oxidase Serum Activity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sciotec Diagnostic Technologies GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BTS1077/17
Record Dates: First submitted 2017-09-26; First posted 2017-10-02 (Actual); Last update posted 2018-04-17 (Actual); Status verified 2017-09

CONDITIONS: Food Intolerance; Histamine Intolerance
Keywords: food intolerance; histamine intolerance; diamine oxidase; DAO; DAOsin
MeSH Terms: conditions — Food Intolerance

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DAOsin treatment (Experimental): Patients suffering from histamine intolerance and a diamin oxidase activity below 10 Units/ml get a DAOsin treatment for one month 3 times a day.
  Interventions: Dietary Supplement: DAOsin

INTERVENTIONS:
Dietary Supplement: DAOsin — DAOsin is a food supplement for special medical purpose for the treatment of food intolerance provoked by histamine intake.

SUMMARY:
DAOsin is a food supplement for special medical purpose for the treatment of food intolerance provoked by histamine intake. In this uncontrolled, interventional pilot study the effect of an oral diamine oxidase substitution (DAOsin) on the reduced endogenous diamine oxidase activity in histamine intolerant patients will be examined.

Patients with a low endogenous diamine oxidase activity (below 10 Units/ml) take DAOsin for one month 3 times a day. During this month the diamine oxidase activity is tested biweekly. Afterwards a follow up period of one month without taking DAOsin follows. Again the diamine oxidase activity is tested biweekly.

ELIGIBILITY:
Inclusion Criteria:

* diamine oxidase activity < 10 U/ml
* >= 2 symptoms of histamine intolerance after consumption of histamine containing food
* 18 to 80 years
* no lactose intolerance
* no fructose intolerance
* no tissue transglutaminase antibodies in serum

Exclusion Criteria:

* pregnancy and nursing
* cardiopathy
* instable hypertonie
* asthma bronchial
* lactose intolerance, fructose intolerance, coeliac disease
* severe liver and kidney diseases
* Known food and other allergies
* participation in clinical study the last 4 weeks
* recent (3 months) operation affecting the gastrointestinal tract
* maligne, infectious or autoimmune gastrointestinal diseases (e.g. IBD)
* taking histamine liberating drugs on a regular basis
* taking diamine oxidase inhibiting drugs on a regular basis
* taking diamine oxidase supplements on a regular basis in the last 4 weeks
* H1 blocker or Montelukast Therapy 4 month before study start
* Taking anti histaminica
* Taking zinc preparations
* drug, alcohol, pharmaceutical abuses
* heavy smoking (>15 cigarettes a day)
* Known HIV infection
* known acute or chronic hepatitis B and C infection

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-08-21 (Actual); Primary Completion 2017-12-06 (Actual); Study Completion 2018-04-16 (Actual)

PRIMARY OUTCOMES:
Change in baseline activity of diamine oxidase activity in serum | 1 month treatment with 1 month follow up
  The activity of diamine oxidase is reduced in patients suffering from histamine intolerance. Supplementation with diamine oxidase helps to reduce the level of histamine coming from food entering the circulation. It is already described that people suffering from histamine intolerance following a histamine reduced diet increase their diamine oxidase activity. The purpose is to test if an additional reduction of probably hidden sources of histamine in food through the administration of DAOsin helps to increase the endogenous diamine oxidase activity even further.

SECONDARY OUTCOMES:
Symptoms of histamine intolerance | 1 month with 1 month follow up
  Every proband documents the severity of histamine intolerance symptoms in a questionnaire.
Histamine level in plasma | 1 month with 1 month follow up
  Is the histamine level in plasma changing upon DAOsin treatment
Global assessment | 1 month with 1 month follow up
  Overall condition during study

CONTACTS AND LOCATIONS:
Locations (1):
- Ordination für Innere Medizin und Stoffwechselzentrum, Bruck an der Mur, Austria

REFERENCES:
- [Derived] Schnedl WJ, Schenk M, Lackner S, Enko D, Mangge H, Forster F. Diamine oxidase supplementation improves symptoms in patients with histamine intolerance. Food Sci Biotechnol. 2019 May 24;28(6):1779-1784. doi: 10.1007/s10068-019-00627-3. eCollection 2019 Dec. PMID 31807350